CLINICAL TRIAL: NCT01169168
Title: Measurement of Fibrinogen in Patients With Systemic Inflammatory Response Syndrome, Sepsis, Chronicle Liver Disease or After Lysis on Intensive Care Units
Brief Title: Measurement of Fibrinogen in Patients With Systemic Inflammatory Response Syndrome (SIRS), Sepsis or Chronicle Liver Disease on Intensive Care Units (ICU)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Dr. med. Wolfgang Miesbach, Johann Wolfgang Goethe University Hospital
Other Study IDs: FibICU
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: SIRS; Sepsis; Liver Disease
Keywords: fibrinogen; SIRS; sepsis; liver disease; chronic liver disease; septic shock
MeSH Terms: conditions — Sepsis; Liver Diseases; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — citrated plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study patients with

1. chronicle liver diseases

   * primary biliary cirrhosis
   * primary sclerosing cholangitis
   * alcoholic liver cirrhosis
   * hepatitis b or C
   * Wilson's disease
   * cryptogenic cirrhosis
2. Septic Inflammatory Response Syndrome (SIRS)

   * sepsis
   * septic shock
3. patients after lysis

should be included

Blood samples will be gathered from the patients to measure fibrinogen with 5 different methods.

The methods are:

* Clauss fibrinogen
* PT-Derived fibrinogen
* immunoturbidimetric method
* heat-precipitated fibrinogen
* Schulz fibrinogen

The result of these tests will be correlated with laboratory values which are gathered in routine and the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* SIRS
* sepsis
* septic shock
* chronicle liver disease (MELD-Score >10)
* patient after lysis
* patient agrees

Exclusion Criteria:

* no agreement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in intensive care units of the university hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-04

PRIMARY OUTCOMES:
Fibrinogen levels from 5 test methods
  * Clauss fibrinogen
  * PT-Derived fibrinogen
  * immunoturbidimetric method
  * heat-precipitated fibrinogen
  * Schulz fibrinogen

SECONDARY OUTCOMES:
Number of bleedings
Number of administered fresh frozen plasma
Number of administered erythrocyte concentrates
Number of administered thrombocyte concentrates
mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Hesse, Germany